CLINICAL TRIAL: NCT04486846
Title: Evaluation of an Electronic Post-Treatment Surveillance Program for Prostate Cancer Survivors (eHealth)
Brief Title: Electronic Post-Treatment Surveillance Program for Prostate Cancer Survivors (eHealth)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left Duke University
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00104751
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eVisit (Experimental): The study intervention will be an electronically performed surveillance program replacing face-to-face clinic follow-up visits. At 3 month intervals for 1 year, the patient will receive an email reminder generated by the patient portal to complete lab testing and eVisit questionnaire.
  Interventions: Other: eVisit

INTERVENTIONS:
Other: eVisit — electronic surveillance program in lieu of in-person clinic visit

SUMMARY:
The purpose of this single institution pilot study is to determine the feasibility of implementing an eHealth prostate cancer surveillance program through the eVisit electronic medical record patient portal. The investigators will assess patient compliance and satisfaction with eVisit follow up care in lieu of in person clinic visits.

DETAILED DESCRIPTION:
Telehealth offers the opportunity to transform cancer surveillance into a patient-centered effort with shared leadership between patient and oncologist. Peer-to-peer electronic communications can improve the collaboration between oncologist and primary care provider (PCP) as patients transition back to primary care as their primary health provider. The investigators propose to test a patient-centered eHealth surveillance program utilizing novel asynchronous telehealth tools to provide patient-reported outcome symptom monitoring using the electronic medical record's patient portal (eVisit).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old with histologically confirmed prostate cancer
* Completed curative intent treatment to the prostate +/- pelvis
* Deemed to be "without evidence of active disease" by treating provider with at least 1 follow up visit 3 or more months after treatment completion
* MyChart account or willingness to open account
* Access to the internet

Exclusion Criteria:

* Documented extrapelvic metastases
* PSA meeting definition of recurrence (>0.2 ng/ml for prostatectomy patients or nadir + 2 ng/ml for radiation patients) and rising with doubling time less than 1 year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete all scheduled eVisits at the end of follow-up | 12 months
  Defined as completion of labwork and at least 80% of the questions asked at each eVisit

SECONDARY OUTCOMES:
Feasibility of enrollment to the eVisit program | 12 months
  Defined as the percentage of patients who are approached for eVisit and ultimately enroll
eVisit participant reported satisfaction | 12 months
  Reported as the summary score from validated Brief Patient Satisfaction 10-item scale instrument assessed from "1/strongly agree" through "5/strongly disagree"
Number of participants with cancer treatment related toxicities | 12 months
  Defined specifically as CTCAE Grade 2 or higher GI, GU, hormonal, and sexual toxicities
Number of eVisit participants with cancer recurrence | 12 months
  Defined as biochemical progression (PSA >0.2 ng/ml for prostatectomy patients or nadir + 2 ng/ml for radiation patients) or metastasis (by imaging)
Financial impact of the eVisit program on participants compared to in person follow up clinic visits | 12 months
  Defined by the financial burden assessment completed by participants, scored from "0/not at all" through "4/very much"
Financial impact of the eVisit program on Duke University Hospital (institution) compared to in person follow up | 12 months
  Defined by percentage of participants/eVisits covered by insurance
Financial impact of the eVisit program on Duke University Hospital (institution) compared to in person follow up | 12 months
  Defined by qualitative analysis of time commitment for providers
Financial impact of the eVisit program on Duke University Hospital (institution) compared to in person follow up | 12 months
  Defined by qualitative analysis of reimbursement process

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Koontz, MD, Principal Investigator — Duke Health
Locations (4):
- United States (4):
  - Duke Cancer Institute Cary, Cary, North Carolina
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No